CLINICAL TRIAL: NCT04634409
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Mono and Combination Therapy With Monoclonal Antibodies in Participants With Mild to Moderate COVID-19 Illness (BLAZE-4)
Brief Title: A Study of Immune System Proteins in Participants With Mild to Moderate COVID-19 Illness
Acronym: BLAZE-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AbCellera Biologics Inc. (Industry); Shanghai Junshi Bioscience Co., Ltd. (Other); GlaxoSmithKline (Industry); Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18160; J2X-MC-PYAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; etesevimab; sotrovimab; bebtelovimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Includes open label arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Pbo) (Placebo Comparator): Treatment 1: Pbo administered intravenously (IV).
  Treatment 8: Pbo For 700 mg Bamlanivimab (BAM) + 500 mg VIR-7831 (Amendment (C-e)) administered IV.
  Treatment 11: Pbo For 175 mg Bebtelovimab (BEB) & 700 mg BAM +1400 mg Etesevimab ( ETE) +175 mg BEB (Low Risk Participants) administered IV.
  Pooled Placebo (Addendum 4, IV) administered IV.
  Pooled Placebo (Addendum 4, SC) administered SC.
  Interventions: Drug: Placebo
- BAM + ETE (Experimental): Treatment 2: 175 mg BAM +350 mg ETE administered IV.
  Treatment 3: 700 mg BAM +1400 mg ETE administered IV.
  Treatment 4: 2800 mg BAM +2800 mg ETE administered IV.
  Treatment 6: 350 mg BAM +700 mg ETE administered IV.
  Unintentional Dosing: 700 mg BAM +700 mg ETE administered IV.
  700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) administered IV.
  700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) administered IV.
  Interventions: Drug: Bamlanivimab; Drug: Etesevimab
- BAM (Experimental): Treatment 5: 700 mg BAM administered IV.
  700 mg BAM 15-min (Addendum (2)) administered IV.
  Interventions: Drug: Bamlanivimab
- BAM + VIR-7831 (Experimental): Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) administered IV.
  Interventions: Drug: Bamlanivimab; Drug: VIR-7831
- BEB (Experimental): Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) administered IV.
  Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) administered IV.
  70 mg BEB 140 mg/Min (Addendum 4, IV) administered IV.
  175 mg BEB 140 mg/Min (Addendum 4, IV) administered IV.
  175 mg BEB 350 mg/Min (Addendum 4, IV) administered IV.
  1750 mg BEB 350 mg/Min (Addendum 4, IV) administered IV.
  280 mg BEB (Addendum 4, SC) administered SC.
  560 mg BEB (Addendum 4, SC) administered SC.
  Interventions: Drug: Bebtelovimab
- BAM+ ETE + BEB (Experimental): Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) administered IV.
  Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) administered IV.
  Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk, Updated Centers for Disease Control and Prevention (CDC) Criteria) administered IV.
  175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) administered IV.
  Interventions: Drug: Bamlanivimab; Drug: Etesevimab; Drug: Bebtelovimab

INTERVENTIONS:
Drug: Bamlanivimab — Administered IV.
  Other Names: LY-CoV555; LY3819253
  Arms: BAM; BAM + ETE; BAM + VIR-7831; BAM+ ETE + BEB
Drug: Etesevimab — Administered IV.
  Other Names: LY-CoV016; LY3832479
  Arms: BAM + ETE; BAM+ ETE + BEB
Drug: Placebo — Administered IV.
  Arms: Placebo (Pbo)
Drug: VIR-7831 — Administered IV.
  Other Names: GSK4182136
  Arms: BAM + VIR-7831
Drug: Bebtelovimab — Administered IV.
  Other Names: LY-CoV1404, LY3853113
  Arms: BAM+ ETE + BEB; BEB

SUMMARY:
The purpose of this study is to measure how well monoclonal antibodies work, either alone or in combination, against the virus that causes COVID-19. Study drug(s) will be given to participants with early symptoms of COVID-19. Samples will be taken from the back of the nose to determine how much virus is in the body at various times during the study. Participation could last about 12 or 24 weeks and includes at least 1 visit to the study site, with the remainder of assessments performed in the home, local clinic, or by phone.

ELIGIBILITY:
Inclusion Criteria:

* For low-risk participant arms 9-11 only: Are greater than or equal to (≥)18 and less than (<)65 years of age at the time of randomization and do not have the risk factors defined in the bullet point directly below
* For high-risk participant arms 12 and 13 only:

  -- Are ≥18 years of age and satisfy at least one of the following risk factors at the time of screening
  * Are ≥65 years of age
  * Have a body mass index (BMI) ≥ 35
  * Have chronic kidney disease
  * Have type 1 or type 2 diabetes
  * Have immunosuppressive disease
  * Are currently receiving immunosuppressive treatment, or
  * Are ≥55 years of age AND have

    * cardiovascular disease, OR
    * hypertension, OR
    * chronic obstructive pulmonary disease or other chronic respiratory disease
* For high-risk participant arms 12 and 13 only:

  * Are 12-17 years of age (inclusive) AND satisfy at least one of the following risk factors at the time of screening

    * Have a BMI ≥85th percentile for their age and gender based on CDC growth charts, https://www.cdc.gov/growthcharts/clinical_charts.htm
    * Have sickle cell disease
    * Have congenital or acquired heart disease
    * Have neurodevelopmental disorders, for example, cerebral palsy
    * Have a medical-related technological dependence, for example, tracheostomy, gastrostomy, or positive pressure ventilation (not related to COVID-19)
    * Have asthma or reactive airway or other chronic respiratory disease that requires daily medication for control
    * Have type 1 or type 2 diabetes
    * Have chronic kidney disease
    * Have immunosuppressive disease, or
    * Are currently receiving immunosuppressive treatment.

For high-risk participants arm 14 only:

* Are ≥12 years of age and satisfy at least one of the following risk factors at the time of screening Are ≥65 years of age
* Are adults (≥18 years of age) with BMI >25 kg/m2 , or if age 12-17, have BMI ≥85th percentile for their age and gender based on CDC growth charts
* Have chronic kidney disease
* Have type 1 or type 2 diabetes
* Have immunosuppressive disease
* Are currently receiving immunosuppressive treatment
* Have cardiovascular disease (including congenital heart disease) or hypertension
* Have chronic lung diseases (for example, chronic obstructive pulmonary disease, asthma [moderate-to-severe], interstitial lung disease, cystic fibrosis and pulmonary hypertension)
* Have sickle cell disease
* Have neurodevelopmental disorder (for example, cerebral palsy) or other conditions that confer medical complexity (for example, genetic or metabolic syndromes and severe congenital anomalies)
* Have a medical-related technological dependence (for example, tracheostomy, gastrostomy, or positive pressure ventilation [not related to COVID-19]
* Are currently not hospitalized
* Have one or more mild or moderate COVID-19 symptoms: Fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, or shortness of breath with exertion, nasal congestion or runny nose, new loss of smell, chills
* Must have sample taken for test confirming viral infection no more than 3 days prior to starting the drug infusion
* Are men or non-pregnant women who agree to contraceptive requirements
* Understand and agree to comply with planned study procedures
* Agree to the collection of nasopharyngeal swabs and venous blood
* The participant or legally authorized representative give signed informed consent and/or assent

Exclusion Criteria:

* For low-risk participants only: BMI ≥35
* Have oxygen saturation (SpO2) less than or equal to (≤)93 percent (%) on room air at sea level or ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) <300, respiratory rate ≥30 per minute, heart rate ≥125 per minute
* Require mechanical ventilation or anticipated impending need for mechanical ventilation
* Have known allergies to any of the components used in the formulation of the interventions
* Have hemodynamic instability requiring use of pressors within 24 hours of randomization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
* Have any co-morbidity requiring surgery within <7 days, or that is considered life-threatening within 29 days
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study
* Have a history of a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test prior to the one serving as eligibility for this study
* Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing
* Have received treatment with a SARS-CoV-2 specific monoclonal antibody
* Have a history of convalescent COVID-19 plasma treatment
* For low-risk arms only: have received a SARS-CoV-2 vaccine or have participated in a previous SARS-CoV-2 vaccine study and are currently blinded to treatment allotment
* Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed
* Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are pregnant or breast feeding
* Are investigator site personnel directly affiliated with this study
* Have body weight <40 kilograms

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1755 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (141):
- United States (127):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Institute for Liver Health, Mesa, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - CRI of Arizona, LLC, Sun City West, Arizona
  - Fiel Family and Sports Medicine PC, Tempe, Arizona
  - The Institute for Liver Health, Tucson, Arizona
  - KLR Business Group, Inc. dba Arkansas Clinical Research, Little Rock, Arkansas
  - Applied Rsch Ctr - Arkansas Inc., Little Rock, Arkansas
  - Smart Cures Clin Research, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - VCT-Covina, Covina, California
  - Neighborhood Healthcare, Escondido, California
  - Chemidox Clinical Trials, Lancaster, California
  - Ark Clinical Research, Long Beach, California
  - Long Beach Clinical Trials LLC, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Central Valley Research, LLC, Modesto, California
  - Inland Empire Liver Foundation, Rialto, California
  - Sutter Institute For Medical Research, Sacramento, California
  - Wolverine Clinical Trials, LLC, Santa Ana, California
  - St. Joe Heritage HC-Santa Rosa, Santa Rosa, California
  - Stanford University Hospital, Stanford, California
  - Mazur, Statner, Dutta, Nathan, Thousand Oaks, California
  - South Bay Clinical Research Institute, Torrance, California
  - Infect Disease Doctors Med Grp, Walnut Creek, California
  - Allianz Research Institute, Westminster, California
  - Future Innovative Treatments LLC, Colorado Springs, Colorado
  - Georgetown Univ Sch of Med, Washington D.C., District of Columbia
  - Synergy Healthcare LLC, Bradenton, Florida
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - I R & Health Center, Inc., Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - Elixia CRC, Hollywood, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Hope Clinical Trials, Inc., Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Clinical Site Partners, LLC d/b/a CSP Miami, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Testing Matters Lab, Sunrise, Florida
  - Advent Health Tampa, Tampa, Florida
  - Triple O Research Inst, West Palm Beach, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Clinical Site Partners, LLC DBA CSP Orlando, Winter Park, Florida
  - Gwinnett Research Inst, Buford, Georgia
  - Paramount Rch Sol - College Pk, College Park, Georgia
  - IACT Health - VHC, Columbus, Georgia
  - Central Georgia Infectious Disease, Macon, Georgia
  - Rophe Adult and Pediatric Medicine, Union City, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Franciscan Health Hammond, Dyer, Indiana
  - Qualmedica Research Evansville, Evansville, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - St.Vincent - Indy, Indianapolis, Indiana
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Tandem Clinical Research,LLC, Marrero, Louisiana
  - Imperial Health Urgent Care Center - Moss Bluff, Moss Bluff, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - U of MA Mem Med Ctr, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Revival Research Institute, Sterling Heights, Michigan
  - Sky Clinical Prime and Health Wellness Clinic, Fayette, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Sky Clin Resch - Quinn HC, Ridgeland, Mississippi
  - Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - SVG Clinical, Las Vegas, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - Prime Global Research, LLC, The Bronx, New York
  - Onsite Clinical Solutions, LLC, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Monroe Biomed Research, Monroe, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Hometown UC and Rch- Cincy, Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Urgent Care Specialists, LLC, Columbus, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - Urgent Care Specialists, LLC, Dayton, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Ascension St. John Tulsa OK, Tulsa, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson Hosp for Neurosci, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - VITALINK - Anderson, Anderson, South Carolina
  - Carolina Medical Research - Clinton, Clinton, South Carolina
  - VITALINK - Gaffney, Gaffney, South Carolina
  - Carolina Medical Research - Greenville, Greenville, South Carolina
  - VITALINK - Greenville, Greenville, South Carolina
  - VITALINK - Spartanburg, Spartanburg, South Carolina
  - VITALINK - Union, Union, South Carolina
  - Univ Diab & Endo Consult, Chattanooga, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Gadolin Research, LLC, Beaumont, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - Crossroads Clinical Research, Corpus Christi, Texas
  - B S & W Med Center, Dallas, Texas
  - Baylor - Fort Worth, Fort Worth, Texas
  - North Texas Clinical Trials, LLC, Fort Worth, Texas
  - Houston Methodist Research Ins, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - Accurate Clinical Management, LLC., Houston, Texas
  - 1960 Family Practice, PA, Houston, Texas
  - B S & W Med Center, Irving, Texas
  - Zion Urgent Care Clinic, Katy, Texas
  - BioPharma Family Practice Center McAllen, McAllen, Texas
  - BRCR Medical Center, Inc, McAllen, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - Bay Area Infectious Diseases Associates, Pasadena, Texas
  - Epic Medical Research, Red Oak, Texas
  - Baylor - Round Rock, Round Rock, Texas
  - Sun Research Institute, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - APD Clinical Research, Splendora, Texas
  - Crossroads Clin Rch-Victoria, Victoria, Texas
  - CLS Research Ctr, PLLC, Webster, Texas
  - CARE ID, Annandale, Virginia
  - Evergreen Health Research, Kirkland, Washington
- Argentina (11):
  - Sanatorio Sagrado Corazón, Ciudad de Buenos Aires, AR
  - Clínica Zabala, Ciudad de Buenos Aires, AR
  - Sanatorio de la Trinidad Mitre, CABA, Buenos Aires
  - Clínica Privada Independencia, Munro, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Instituto Médico Rio Cuarto, Río Cuarto, Córdoba Province
  - Centro de Investigaciones Clínicas - Clínica Viedma, Viedma, Río Negro Province
  - Clinica Central S.A., Villa Regina, Río Negro Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Hospital San Roque, Córdoba
- Puerto Rico (3):
  - Advanced Clinical Research, LLC, Bayamón
  - Dorado Medical Complex Inc, Dorado
  - GCM Medical Group, PSC - Hato Rey Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
URL: http://vivli.org/

REFERENCES:
- [Derived] Nichols RM, Macpherson L, Patel DR, Yeh WW, Peppercorn A. Effect of Bamlanivimab as Monotherapy or in Combination with Etesevimab or Sotrovimab on Persistently High Viral Load in Patients with Mild-to-Moderate COVID-19: A Randomized, Phase 2 BLAZE-4 Trial. Infect Dis Ther. 2024 Feb;13(2):401-411. doi: 10.1007/s40121-024-00918-1. Epub 2024 Jan 30. PMID 38291279
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Nathan R, Shawa I, De La Torre I, Pustizzi JM, Haustrup N, Patel DR, Huhn G. A Narrative Review of the Clinical Practicalities of Bamlanivimab and Etesevimab Antibody Therapies for SARS-CoV-2. Infect Dis Ther. 2021 Dec;10(4):1933-1947. doi: 10.1007/s40121-021-00515-6. Epub 2021 Aug 10. PMID 34374951
- See also: A Study of Immune System Proteins in Participants With Mild to Moderate COVID-19 Illness — https://trials.lillytrialguide.com/en-US/trial/3GPxb8Mwm9PjgI7IrKcsTB

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1: Pbo: Participants received placebo (Pbo) administered intravenously (IV).
- Treatment 2: 175 mg BAM +350 mg ETE: Participants received 175 milligrams (mg) bamlanivimab (BAM) +350 mg etesevimab (ETE) administered IV.
- Treatment 3: 700 mg BAM +1400 mg ETE: Participants received 700 mg BAM +1400 mg ETE administered IV.
- Treatment 4: 2800 mg BAM +2800 mg ETE: Participants received 2800 mg BAM + 2800 mg ETE administered IV.
- Treatment 5: 700 mg BAM: Participants received 700 mg BAM administered IV.
- Treatment 6: 350 mg BAM +700 mg ETE: Participants received 350 mg BAM +700 mg ETE administered IV.
- Unintentional Dosing: 700 mg BAM +700 mg ETE: Participants received 700 mg BAM +700 mg ETE administered IV.
- Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)): Participants received 700 mg BAM + 500 mg VIR-7831 administered IV.
- Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)); Pooled Placebo (Addendum 4, IV): Participants received placebo administered IV.
- Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants): Amendment (f) Low Risk Participants:
  Participants received 175 mg bebtelovimab (BEB) administered IV.
- Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants): Amendment (f) Low Risk Participants:
  Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV.
- Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants): Amendment (f) Low Risk Participants:
  Participants received placebo administered IV.
- Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants): Amendment (f) High Risk Participants:
  Participants received 175 mg BEB administered IV.
- Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants): Amendment (f) High Risk Participants:
  Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV.
- Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria): Amendment (g), High Risk, Updated CDC Criteria):
  Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV for participants in updated CDC criteria.
- 700 mg BAM 15-min (Addendum (2)): Participants received 700 mg BAM administered IV.
  Addendum 2 explored the safety of accelerated intravenous (IV) administration of BAM alone and in combination with ETE.
- 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)); 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)): Participants received 700 mg BAM +1400 mg ETE administered IV.
  Addendum 2 explored the safety of accelerated intravenous (IV) administration of BAM alone and in combination with ETE.
- 70 mg BEB 140 mg/Min (Addendum 4, IV): Participants received 70 mg BEB 140 mg/min IV.
- 175 mg BEB 140 mg/Min (Addendum 4, IV): Participants received 175 mg BEB 140 mg/min IV.
- 175 mg BEB 350 mg/Min (Addendum 4, IV): Participants received 175 mg BEB 350 mg/min IV.
- 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV): Participants received 175 mg BAM + 700 mg ETE + 1400 mg BEB 350 mg/min IV.
- 1750 mg BEB 350 mg/Min (Addendum 4, IV): Participants received 1750 mg BEB 350 mg/min IV.
- Pooled Placebo (Addendum 4, SC): Participants received Placebo SC.
- 280 mg BEB (Addendum 4, SC): Participants received 280 mg BEB SC.
- 560 mg BEB (Addendum 4, SC): Participants received 560 mg BEB SC.
Period: Overall Study
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg BAM +700 mg ETE | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria) | 700 mg BAM 15-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) | Pooled Placebo (Addendum 4, IV) | 70 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 350 mg/Min (Addendum 4, IV) | 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) | 1750 mg BEB 350 mg/Min (Addendum 4, IV) | Pooled Placebo (Addendum 4, SC) | 280 mg BEB (Addendum 4, SC) | 560 mg BEB (Addendum 4, SC)
Started | 155 | 83 | 158 | 103 | 105 | 101 | 20 (During the study period, 20 participants from the BAM 175-mg + ETE 350-mg arm potentially received 700 mg bamlanivimab + 700 mg etesevimab instead. These 20 participants, who were randomized at 8 different sites were identified through pharmacokinetics analyses.) | 101 | 101 | 125 | 127 | 128 | 100 | 50 | 176 | 30 | 6 | 30 | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Received at Least One Dose of Study Drug | 155 | 83 | 158 | 103 | 105 | 101 | 20 | 101 | 101 | 125 | 127 | 128 | 100 | 50 | 176 | 30 | 6 | 30 | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Completed | 148 | 81 | 150 | 96 | 102 | 99 | 19 | 90 | 91 | 112 | 114 | 109 | 92 | 46 | 164 | 30 | 6 | 29 | 10 | 6 | 6 | 6 | 6 | 5 | 4 | 6 | 6
Not Completed | 7 | 2 | 8 | 7 | 3 | 2 | 1 | 11 | 10 | 13 | 13 | 19 | 8 | 4 | 12 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 1 | 3 | 1 | 1 | 1 | 3 | 3 | 11 | 8 | 15 | 3 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 6 | 4 | 2 | 0 | 0 | 2 | 3 | 2 | 3 | 2 | 2 | 1 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other - As reported by Investigator | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab: Participants received 700 mg bamlanivimab +700 mg etesevimab administered IV.
- Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants): Amendment (f) Low Risk Participants:
  Participants received 175 mg BEB administered IV.
- Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g), Updated CDC Criteria): Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV for participants in updated CDC criteria.
- 280 BEB (Addendum 4, SC): Participants received 280 mg BEB SC.
- Total: Total of all reporting groups
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g), Updated CDC Criteria) | 700 mg BAM 15-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) | Pooled Placebo (Addendum 4, IV) | 70 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 350 mg/Min (Addendum 4, IV) | 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) | 1750 mg BEB 350 mg/Min (Addendum 4, IV) | Pooled Placebo (Addendum 4, SC) | 280 BEB (Addendum 4, SC) | 560 mg BEB (Addendum 4, SC) | Total
Number analyzed (Participants) | 155 | 83 | 158 | 103 | 105 | 101 | 20 | 101 | 101 | 125 | 127 | 128 | 100 | 50 | 176 | 30 | 6 | 30 | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 1755
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.22) | 41.5 (12.89) | 37.7 (12.11) | 39.5 (12.63) | 39.8 (12.70) | 42.3 (11.93) | 36.5 (15.04) | 37.6 (12.83) | 38.9 (11.77) | 36.2 (11.40) | 37.6 (12.12) | 36.1 (11.66) | 49.1 (15.17) | 50.8 (17.06) | 49.3 (17.39) | 35.4 (12.55) | 47.7 (7.28) | 42.9 (11.87) | 46.8 (13.27) | 35.2 (13.99) | 48.7 (9.83) | 36.3 (15.24) | 41.7 (14.76) | 39.5 (16.88) | 30.0 (6.98) | 35.8 (7.08) | 39.2 (9.70) | 40.6 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 39 | 86 | 55 | 50 | 48 | 8 | 52 | 56 | 63 | 76 | 72 | 52 | 26 | 98 | 12 | 3 | 13 | 3 | 3 | 6 | 1 | 3 | 5 | 1 | 1 | 2 | 909
  Male | 80 | 44 | 72 | 48 | 55 | 53 | 12 | 49 | 45 | 62 | 51 | 56 | 48 | 24 | 78 | 18 | 3 | 17 | 7 | 3 | 0 | 5 | 3 | 1 | 3 | 5 | 4 | 846
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 24 | 47 | 28 | 28 | 33 | 3 | 18 | 27 | 46 | 45 | 45 | 19 | 8 | 49 | 15 | 1 | 3 | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 497
  Not Hispanic or Latino | 104 | 57 | 108 | 70 | 74 | 66 | 17 | 80 | 72 | 78 | 82 | 83 | 81 | 42 | 126 | 15 | 5 | 26 | 6 | 6 | 6 | 5 | 5 | 4 | 4 | 2 | 4 | 1228
  Unknown or Not Reported | 3 | 2 | 3 | 5 | 3 | 2 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13
  Asian | 4 | 4 | 13 | 3 | 9 | 4 | 0 | 4 | 1 | 1 | 4 | 2 | 3 | 1 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Black or African American | 7 | 5 | 6 | 7 | 4 | 7 | 2 | 15 | 5 | 19 | 19 | 29 | 14 | 13 | 28 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 185
  White | 132 | 68 | 127 | 91 | 85 | 84 | 17 | 74 | 90 | 97 | 99 | 90 | 78 | 32 | 136 | 27 | 3 | 27 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 1410
  More than one race | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Unknown or Not Reported | 9 | 6 | 7 | 2 | 5 | 5 | 1 | 4 | 4 | 8 | 5 | 6 | 0 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 155 | 83 | 158 | 103 | 105 | 101 | 20 | 101 | 101 | 125 | 127 | 128 | 100 | 50 | 176 | 30 | 6 | 30 | 10 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 1755

OUTCOME MEASURES:

1. Primary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Percentage of Participants With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load Greater Than 5.27
Description: Percentage of participants with SARS-CoV-2 viral load greater than 5.27 on Day 7. Missing data is estimated using Relevance Sequence Imputation (RSI). RSI is defined as follows: If Day 7 SARS-CoV-2 viral load is missing, then Day 7 will be imputed using data from the first available for Day 5, Day 3, Day 11, or Day 1.
Time Frame: Day 7
Population: Treatment 1-6 and Unintentional Dosing arms: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg BAM +700 mg ETE
Number analyzed (Participants) | 155 | 82 | 157 | 103 | 105 | 101 | 20
percentage of participants | 27.7 [20.7 to 34.8] | 12.2 [5.1 to 19.3] | 10.8 [6.0 to 15.7] | 7.8 [2.6 to 12.9] | 14.3 [7.6 to 21.0] | 7.9 [2.7 to 13.2] | 10.0 [0.0 to 23.1]
Statistical Analysis 1: Comparison: Treatment 1: Pbo vs Treatment 2: 175 mg BAM +350 mg ETE; Test type: Superiority; p = 0.009273, Regression, Logistic; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.18 to 0.78]
Statistical Analysis 2: Comparison: Treatment 1: Pbo vs Treatment 3: 700 mg BAM +1400 mg ETE; Test type: Superiority; p = 0.000271, Regression, Logistic; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.18 to 0.59]
Statistical Analysis 3: Comparison: Treatment 1: Pbo vs Treatment 4: 2800 mg BAM +2800 mg ETE; Test type: Superiority; p = 0.000257, Regression, Logistic; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.10 to 0.51]
Statistical Analysis 4: Comparison: Treatment 1: Pbo vs Treatment 5: 700 mg BAM; Test type: Superiority; p = 0.013378, Regression, Logistic; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.23 to 0.84]
Statistical Analysis 5: Comparison: Treatment 1: Pbo vs Treatment 6: 350 mg BAM +700 mg ETE; Test type: Superiority; p = 0.000318, Regression, Logistic; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.11 to 0.52]
Statistical Analysis 6: Comparison: Treatment 1: Pbo vs Unintentional Dosing: 700 mg BAM +700 mg ETE; Test type: Superiority; p = 0.140563, Regression, Logistic; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.09 to 1.41]

2. Primary Outcome: Treatment 7-8, Amendments (C-e): Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: Percentage of participants with SARS-CoV-2 viral load greater than 5.27 on Day 7. Missing data is estimated using Last Observation Carried Forward (LOCF).
Time Frame: Day 7
Population: Treatment 7-8, Amendments (C-e): All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 101 | 101
percentage of participants | 9.9 [4.1 to 15.7] | 29.7 [20.8 to 38.6]
Statistical Analysis 1: Comparison: Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) vs Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)); Test type: Superiority; p = 0.000835, Regression, Logistic; Odds Ratio (OR) = 0.27, 95% CI 2-sided [0.12 to 0.58]

3. Primary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: as for outcome 2
Time Frame: Day 7
Population: Treatment 9-11 Amendment (f), Low Risk Participants: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants)
Number analyzed (Participants) | 125 | 126 | 126
percentage of participants | 12.0 [6.3 to 17.7] | 12.7 [6.9 to 18.5] | 19.8 [12.9 to 26.8]
Statistical Analysis 1: Comparison: Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.097231, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.28 to 1.11]
Statistical Analysis 2: Comparison: Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.132360, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.30 to 1.17]

4. Secondary Outcome: Treatment 12 -13, Amendment (f) High Risk Participants: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: as for outcome 2
Time Frame: Day 7
Population: Treatment 12 -13, Amendment (f) High Risk Participants: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 99 | 50
percentage of participants | 25.3 [16.7 to 33.8] | 12.0 [3.0 to 21.0]

5. Secondary Outcome: Treatment 14, Amendment (f) High Risk Participants Updated CDC Criteria: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: as for outcome 2
Time Frame: Day 7
Population: Treatment 14, Amendment (f) High Risk Participants Updated CDC Criteria: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria)
Number analyzed (Participants) | 176
percentage of participants | 17.6 [12.0 to 23.2]

6. Secondary Outcome: Addendum (2): Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: Missing data is estimated using Relevance Sequence Imputation (RSI). RSI is defined as follows: If Day 7 SARS-CoV-2 viral load is missing, then Day 7 will be imputed using data from the first available for Day 5, Day 3, Day 11, or Day 1.
Time Frame: Day 7
Population: Addendum (2): All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 700 mg BAM 15-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2))
Number analyzed (Participants) | 30 | 6 | 30
percentage of participants | 16.7 [3.3 to 30.0] | 0.0 [0.0 to 0.0] | 13.3 [1.2 to 25.5]

7. Secondary Outcome: Addendum (4), Arm A - Intravenous: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: as for outcome 2
Time Frame: Day 7
Population: Addendum (4) Arm A - Intravenous: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 175 BEB 140 mg/Min (Addendum 4, IV): Participants received 175 mg BEB 140 mg/min IV.
- 175 BEB 350 mg/Min (Addendum 4, IV): Participants received 175 mg BEB 350 mg/min IV.
- 175/700/1400 BAM+ETE+BEB 350mg/Min (Addendum 4, IV): Participants received 175 mg BAM + 700 mg ETE + 1400 mg BEB 350 mg/min IV.
- 1750 BEB 350 mg/Min (Addendum 4, IV): Participants received 1750 mg BEB 350 mg/min IV.
Arm/Group | Pooled Placebo (Addendum 4, IV) | 70 mg BEB 140 mg/Min (Addendum 4, IV) | 175 BEB 140 mg/Min (Addendum 4, IV) | 175 BEB 350 mg/Min (Addendum 4, IV) | 175/700/1400 BAM+ETE+BEB 350mg/Min (Addendum 4, IV) | 1750 BEB 350 mg/Min (Addendum 4, IV)
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 40.0 [9.6 to 70.4] | 16.7 [0.0 to 46.5] | 50.0 [10.0 to 90.0] | 0.0 [0.0 to 0.0] | 16.7 [0.0 to 46.5] | 33.3 [0.0 to 71.1]

8. Secondary Outcome: Addendum (4) Arm B - Subcutaneous: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than 5.27
Description: as for outcome 2
Time Frame: Day 7
Population: Addendum (4) Arm B - Subcutaneous: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pooled Placebo (Addendum 4, SC): Participants received placebo administered SC.
Arm/Group | Pooled Placebo (Addendum 4, SC) | 280 mg BEB (Addendum 4, SC) | 560 mg BEB (Addendum 4, SC)
Number analyzed (Participants) | 4 | 6 | 6
percentage of participants | 25.0 [0.0 to 67.4] | 16.7 [0.0 to 46.5] | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death from any Cause
Time Frame: Baseline through Day 29
Population: Treatment 1-6 and Unintentional Dosing arms: All participants randomly assigned and who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab
Number analyzed (Participants) | 155 | 83 | 158 | 103 | 105 | 101 | 20
percentage of participants | 0.6 [0.0 to 1.9] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Treatment 1: Pbo vs Treatment 2: 175 mg BAM +350 mg ETE; Test type: Superiority; p = 0.769, Regression, Logistic; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.02 to 15.57]
Statistical Analysis 2: Comparison: Treatment 1: Pbo vs Treatment 3: 700 mg BAM +1400 mg ETE; Test type: Superiority; p = 0.494, Regression, Logistic; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.01 to 8.12]
Statistical Analysis 3: Comparison: Treatment 1: Pbo vs Treatment 4: 2800 mg BAM +2800 mg ETE; Test type: Superiority; p = 0.671, Regression, Logistic; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.02 to 12.51]
Statistical Analysis 4: Comparison: Treatment 1: Pbo vs Treatment 5: 700 mg BAM; Test type: Superiority; p = 0.663, Regression, Logistic; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.02 to 12.27]
Statistical Analysis 5: Comparison: Treatment 1: Pbo vs Treatment 6: 350 mg BAM +700 mg ETE; Test type: Superiority; p = 0.680, Regression, Logistic; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.02 to 12.76]
Statistical Analysis 6: Comparison: Treatment 1: Pbo vs Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab; Test type: Superiority; p = 0.584, Regression, Logistic; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.09 to 67.88]

10. Secondary Outcome: Treatment 7-8, Amendment (C-E): Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death from Any Cause
Time Frame: Baseline through Day 29
Population: Treatment 7-8, Amendment (C-E): All participants randomly assigned and who received any amount of study drug. No participants met the criteria (duration had to be 24 or more, and had to occur on Day 29 or before)
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Time Frame: Baseline through Day 29
Population: Treatment 9-11 Amendment (f), Low Risk Participants: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants)
Number analyzed (Participants) | 125 | 127 | 128
percentage of participants | 1.6 [0.0 to 3.8] | 2.4 [0.0 to 5.0] | 1.6 [0.0 to 3.7]
Statistical Analysis 1: Comparison: Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.979, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.17 to 6.06]
Statistical Analysis 2: Comparison: Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.675, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.27 to 7.39]

12. Secondary Outcome: Treatment 12 -13 Amendment (f), High Risk Participants: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Time Frame: Baseline through Day 29
Population: Treatment 12 -13 Amendment (f), High Risk Participants: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants: Amendment (f) High Risk Participants:
  Participants received 175 mg BEB administered IV.
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 100 | 50
percentage of participants | 3.0 [0.0 to 6.3] | 4.0 [0.0 to 9.4]

13. Secondary Outcome: Treatment 14 Amendment (f) High Risk Participants, Updated CDC Criteria: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Time Frame: Baseline through Day 29
Population: Treatment 14 Amendment (f) High Risk, Participants Updated CDC Criteria: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g) High Risk,Updated CDC Criteria): Amendment (g), High Risk, Updated CDC Criteria):
  Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV for participants in updated CDC criteria.
Arm/Group | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g) High Risk,Updated CDC Criteria)
Number analyzed (Participants) | 176
percentage of participants | 1.7 [0.0 to 3.6]

14. Secondary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: Least squares mean (LSM) change from baseline was calculated using a mixed model repeating measures (MMRM) that included log base 10 transformed baseline as a covariate, treatment, day, treatment-by-day interaction as fixed effects. Viral load is reported as normalized viral and is unitless.
Time Frame: Baseline, Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: unitless
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab
Number analyzed (Participants) | 135 | 71 | 138 | 92 | 93 | 81 | 17
unitless | -2.87 (0.149) | -3.54 (0.207) | -3.52 (0.148) | -3.13 (0.181) | -3.28 (0.180) | -3.74 (0.191) | -3.51 (0.419)
Statistical Analysis 1: Comparison: Treatment 1: Pbo vs Treatment 2: 175 mg BAM +350 mg ETE; Test type: Superiority; p = 0.009, Mixed Models Analysis; LSM Difference = -0.67, 95% CI 2-sided [-1.17 to -0.17]
Statistical Analysis 2: Comparison: Treatment 1: Pbo vs Treatment 3: 700 mg BAM +1400 mg ETE; Test type: Superiority; p = 0.002, Mixed Models Analysis; LSM Difference = -0.65, 95% CI 2-sided [-1.06 to -0.24]
Statistical Analysis 3: Comparison: Treatment 1: Pbo vs Treatment 4: 2800 mg BAM +2800 mg ETE; Test type: Superiority; p = 0.263, Mixed Models Analysis; LSM Difference = -0.26, 95% CI 2-sided [-0.72 to 0.20]
Statistical Analysis 4: Comparison: Treatment 1: Pbo vs Treatment 5: 700 mg BAM; Test type: Superiority; p = 0.083, Mixed Models Analysis; LSM Difference = -0.41, 95% CI 2-sided [-0.87 to 0.05]
Statistical Analysis 5: Comparison: Treatment 1: Pbo vs Treatment 6: 350 mg BAM +700 mg ETE; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = -0.87, 95% CI 2-sided [-1.35 to -0.40]
Statistical Analysis 6: Comparison: Treatment 1: Pbo vs Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab; Test type: Superiority; p = 0.149, Mixed Models Analysis; LSM Difference = -0.64, 95% CI 2-sided [-1.52 to 0.23]

15. Secondary Outcome: Treatment 7-8 Amendments (C-e): Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: LSM change from baseline was calculated using a MMRM that included log base 10 transformed baseline as a covariate, treatment, day, treatment-by-day interaction as fixed effects. Viral load is reported as normalized viral and is unitless.
Time Frame: Baseline, Day 7
Population: Treatment 7-8 Amendments (c-e): All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Least Squares Mean (Standard Error); unit: unitless
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 96 | 94
unitless | -3.56 (0.182) | -2.74 (0.184)
Statistical Analysis 1: Comparison: Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) vs Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)); Test type: Superiority; p = 0.002, Mixed Models Analysis; LSM Difference = -0.82, 95% CI 2-sided [-1.33 to -0.31]

16. Secondary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: as for outcome 15
Time Frame: Baseline, Day 7
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: unitless
Arm/Group | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants)
Number analyzed (Participants) | 113 | 115 | 113
unitless | -3.77 (0.198) | -4.00 (0.196) | -3.62 (0.198)
Statistical Analysis 1: Comparison: Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.606, Mixed Models Analysis; LSM Difference = -0.14, 95% CI 2-sided [-0.70 to 0.41]
Statistical Analysis 2: Comparison: Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.170, Mixed Models Analysis; LSM Difference = -0.38, 95% CI 2-sided [-0.93 to 0.17]

17. Secondary Outcome: Treatment 12 -13 Amendment (f), High Risk Participants: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: Baseline is defined as the last non-missing assessment recorded on or prior to the date of first study drug injection. Viral load is reported as normalized viral and is unitless.
Time Frame: Baseline, Day 7
Population: Treatment 12 -13 Amendment (f), High Risk Participants: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 88 | 47
unitless | -3.22 (2.585) | -3.43 (2.835)

18. Secondary Outcome: Treatment 14, Amendment (f) High Risk Participants Updated CDC Criteria: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: as for outcome 17
Time Frame: Baseline, Day 7
Population: as for outcome 5
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria)
Number analyzed (Participants) | 157
unitless | -4.00 (2.514)

19. Secondary Outcome: Addendum 4, IV: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: as for outcome 17
Time Frame: Baseline, Day 7
Population: Addendum 4, IV: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Pooled Placebo (Addendum 4, IV) | 70 mg BEB 140 mg/Min (Addendum 4, IV) | 175 BEB 140 mg/Min (Addendum 4, IV) | 175 BEB 350 mg/Min (Addendum 4, IV) | 175/700/1400 BAM+ETE+BEB 350mg/Min (Addendum 4, IV) | 1750 BEB 350 mg/Min (Addendum 4, IV)
Number analyzed (Participants) | 8 | 6 | 5 | 6 | 5 | 5
unitless | -4.27 (3.087) | -4.39 (2.334) | -4.40 (3.188) | -4.49 (1.925) | -6.35 (1.502) | -4.76 (2.217)

20. Secondary Outcome: Addendum 4, SC: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: as for outcome 17
Time Frame: Baseline, Day 7
Population: Addendum 4, SC: All randomized participants who received study drug and provided at least 1 postbaseline measure viral load measurement.
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- 560 mg BEB (Addendum 4, SC: Participants received 560 mg BEB SC.
Arm/Group | Pooled Placebo (Addendum 4, SC) | 280 mg BEB (Addendum 4, SC) | 560 mg BEB (Addendum 4, SC
Number analyzed (Participants) | 3 | 6 | 6
unitless | -3.47 (3.934) | -4.04 (2.114) | -3.40 (1.900)

21. Secondary Outcome: Addendum (2): Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: as for outcome 17
Time Frame: Baseline, Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | 700 mg BAM 15-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2))
Number analyzed (Participants) | 27 | 5 | 25
unitless | -2.65 (2.394) | -4.90 (1.999) | -4.37 (2.128)

22. Secondary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Percentage of Participants Demonstrating Symptom Resolution
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and loss in taste and smell. Each symptom (excluding loss of taste and smell) was scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Loss of taste and smell was scored as Yes (Y) or No (N). Symptom resolution (yes/no) is defined as all symptoms (excluding loss of appetite, taste, and smell) on the symptom questionnaire scored as absent (score of 0). Missing data was imputed using a non-responder imputation.
Time Frame: Day 7
Population: Treatment 1-6 and Unintentional Dosing Arms: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Resolution values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab
Number analyzed (Participants) | 155 | 82 | 157 | 103 | 105 | 101 | 20
percentage of participants | 29.0 [21.9 to 36.2] | 28.0 [18.3 to 37.8] | 36.9 [29.4 to 44.5] | 32.0 [23.0 to 41.1] | 41.0 [31.5 to 50.4] | 32.7 [23.5 to 41.8] | 30.0 [9.9 to 50.1]
Statistical Analysis 1: Comparison: Treatment 1: Pbo vs Treatment 2: 175 mg BAM +350 mg ETE; Test type: Superiority; p = 0.890, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.53 to 1.73]
Statistical Analysis 2: Comparison: Treatment 1: Pbo vs Treatment 3: 700 mg BAM +1400 mg ETE; Test type: Superiority; p = 0.141, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.89 to 2.29]
Statistical Analysis 3: Comparison: Treatment 1: Pbo vs Treatment 4: 2800 mg BAM +2800 mg ETE; Test type: Superiority; p = 0.603, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.67 to 1.98]
Statistical Analysis 4: Comparison: Treatment 1: Pbo vs Treatment 5: 700 mg BAM; Test type: Superiority; p = 0.048, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.00 to 2.84]
Statistical Analysis 5: Comparison: Treatment 1: Pbo vs Treatment 6: 350 mg BAM +700 mg ETE; Test type: Superiority; p = 0.533, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.69 to 2.04]
Statistical Analysis 6: Comparison: Treatment 1: Pbo vs Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab; Test type: Superiority; p = 0.869, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.40 to 2.99]

23. Secondary Outcome: Treatment 7-8 Amendments (C-e): Percentage of Participants Demonstrating Symptom Resolution
Description: as for outcome 22
Time Frame: Day 7
Population: Treatment 7-8 Amendments (c-e): All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Resolution values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 101 | 101
percentage of participants | 35.6 [26.3 to 45.0] | 29.7 [20.8 to 38.6]
Statistical Analysis 1: Comparison: Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) vs Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)); Test type: Superiority; p = 0.374, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.72 to 2.35]

24. Secondary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Percentage of Participants Demonstrating Symptom Resolution
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and loss in taste and smell. Each symptom (excluding loss of taste and smell) was scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Loss of taste and smell was scored as Yes (Y) or No (N). Symptom resolution (yes/no) is defined as a score of 0 for shortness of breath, feeling feverish, body aches and pains, sore throat, chills, and headache, and a score of 0 or 1 for cough and fatigue on the symptom questionnaire. Missing data was imputed using a non-responder imputation.
Time Frame: Day 7
Population: Treatment 9-11 Amendment (f), Low Risk Participants: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Resolution values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants)
Number analyzed (Participants) | 125 | 126 | 126
percentage of participants | 60.0 [51.4 to 68.6] | 50.8 [42.1 to 59.5] | 44.4 [35.8 to 53.1]
Statistical Analysis 1: Comparison: Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.13 to 3.08]
Statistical Analysis 2: Comparison: Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) vs Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants); Test type: Superiority; p = 0.317, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.78 to 2.11]

25. Secondary Outcome: Treatment 12 -13 Amendment (f), High Risk Participants: Percentage of Participants Demonstrating Symptom Resolution
Description: as for outcome 24
Time Frame: Day 7
Population: Treatment 12 -13 Amendment (f), High Risk Participants: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Resolution values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 99 | 50
percentage of participants | 50.5 [40.7 to 60.4] | 52.0 [38.2 to 65.8]

26. Secondary Outcome: Treatment 14, Amendment (g) High Risk Participants Updated CDC Criteria Amendment (g): Percentage of Participants Demonstrating Symptom Resolution
Description: as for outcome 24
Time Frame: Day 7
Population: Treatment 14, Amendment (g) High Risk Participants Updated CDC Criteria Amendment (g): All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Resolution values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g)): Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV.
Arm/Group | 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g))
Number analyzed (Participants) | 176
percentage of participants | 47.2 [39.8 to 54.5]

27. Secondary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Percentage of Participants Demonstrating Symptom Improvement
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and loss in taste and smell. Each symptom (excluding loss of taste and smell) was scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Loss of taste and smell was scored as Yes (Y) or No (N). Symptom improvement (yes/no) is defined as a patient experiencing symptoms on the symptom questionnaire (excluding loss of appetite, taste, and smell) scored as moderate or severe (score of 2 or 3) at baseline are subsequently scored as mild or absent (score of 1 or 0), AND symptoms on the symptom questionnaire scored as mild or absent at baseline are subsequently scored as absent.
Time Frame: Day 7
Population: Treatment 1-6 and Unintentional Dosing Arms: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Improvement values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo administered intravenously (IV).
- 175 mg Bamlanivimab +350 mg Etesevimab: Participants received 175 milligrams (mg) bamlanivimab +350 mg etesevimab administered IV.
- 350 mg Bamlanivimab +700 mg Etesevimab: Participants received 350 mg bamlanivimab +700 mg etesevimab administered IV.
- 700 mg Bamlanivimab +1400 mg Etesevimab: Participants received 700 mg bamlanivimab +1400 mg etesevimab administered IV.
- 2800 mg Bamlanivimab +2800 mg Etesevimab: Participants received 2800 mg bamlanivimab + 2800 mg etesevimab administered IV.
- 700 mg Bamlanivimab: Participants received 700 mg bamlanivimab administered IV.
- Unintentional Dosing Arm: 700 mg Bamlanivimab +700 mg Etesevimab: Participants received 700 mg bamlanivimab +700 mg etesevimab administered IV.
Arm/Group | Placebo | 175 mg Bamlanivimab +350 mg Etesevimab | 350 mg Bamlanivimab +700 mg Etesevimab | 700 mg Bamlanivimab +1400 mg Etesevimab | 2800 mg Bamlanivimab +2800 mg Etesevimab | 700 mg Bamlanivimab | Unintentional Dosing Arm: 700 mg Bamlanivimab +700 mg Etesevimab
Number analyzed (Participants) | 155 | 82 | 101 | 157 | 103 | 105 | 20
percentage of participants | 33.5 [26.1 to 41.8] | 45.1 [34.4 to 55.9] | 48.5 [38.8 to 58.3] | 46.5 [38.7 to 54.3] | 49.5 [39.9 to 59.2] | 52.4 [42.8 to 61.9] | 40.0 [18.5 to 61.5]
Statistical Analysis 1: Comparison: Placebo vs 175 mg Bamlanivimab +350 mg Etesevimab; Test type: Superiority; p = 0.082, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.94 to 2.81]
Statistical Analysis 2: Comparison: Placebo vs 350 mg Bamlanivimab +700 mg Etesevimab; Test type: Superiority; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.11 to 3.11]
Statistical Analysis 3: Comparison: Placebo vs 700 mg Bamlanivimab +1400 mg Etesevimab; Test type: Superiority; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.09 to 2.71]
Statistical Analysis 4: Comparison: Placebo vs 2800 mg Bamlanivimab +2800 mg Etesevimab; Test type: Superiority; p = 0.011, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.16 to 3.22]
Statistical Analysis 5: Comparison: Placebo vs 700 mg Bamlanivimab; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.30 to 3.60]
Statistical Analysis 6: Comparison: Placebo vs Unintentional Dosing Arm: 700 mg Bamlanivimab +700 mg Etesevimab; Test type: Superiority; p = 0.546, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.52 to 3.48]

28. Secondary Outcome: Treatment 7-8 Amendments (C-E): Percentage of Participants Demonstrating Symptom Improvement
Description: as for outcome 27
Time Frame: Day 7
Population: Treatment 7-8 Amendments (C-E): All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Improvement values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 101 | 101
percentage of participants | 43.6 [33.9 to 53.2] | 42.6 [32.9 to 52.2]
Statistical Analysis 1: Comparison: Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) vs Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)); Test type: Superiority; p = 0.888, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.60 to 1.82]

29. Secondary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Percentage of Participants Demonstrating Symptom Improvement
Description: as for outcome 27
Time Frame: Day 7
Population: Treatment 9-11 Amendment (f), Low Risk Participants: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and and had non-missing Symptom Improvement values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants)
Number analyzed (Participants) | 126 | 125 | 126
percentage of participants | 34.9 [26.6 to 43.2] | 50.4 [41.6 to 59.2] | 46.8 [38.1 to 55.5]
Statistical Analysis 1: Comparison: Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) vs Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants); Test type: Superiority; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.13 to 3.13]
Statistical Analysis 2: Comparison: Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) vs Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants); Test type: Superiority; p = 0.057, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.98 to 2.71]

30. Secondary Outcome: Treatment 12 -13 Amendment (f), High Risk Participants: Percentage of Participants Demonstrating Symptom Improvement
Description: as for outcome 27
Time Frame: Day 7
Population: Treatment 12 -13 Amendment (f), High Risk Participants: All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Improvement values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 99 | 50
percentage of participants | 42.4 [32.7 to 52.2] | 42.0 [28.3 to 55.7]

31. Secondary Outcome: Treatment 14 Amendment (g): Percentage of Participants Demonstrating Symptom Improvement
Description: as for outcome 27
Time Frame: Day 7
Population: Treatment 14 Amendment (g): All randomized participants who received study drug, provided at least 1 postbaseline measure viral load measurement and had non-missing Symptom Improvement values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria)
Number analyzed (Participants) | 176
percentage of participants | 38.6 [31.4 to 45.8]

32. Secondary Outcome: Treatment 1-6 and Unintentional Dosing Arms: Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Time Frame: Baseline through Day 29
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg Bamlanivimab +700 mg Etesevimab
Number analyzed (Participants) | 155 | 83 | 158 | 103 | 105 | 101 | 20
percentage of participants | 1.9 [0.0 to 4.1] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 1.0 [0.0 to 2.8] | 0.0 [0.0 to 0.0] | 5.0 [0.0 to 14.6]

33. Secondary Outcome: Treatment 7-8 Amendments (C-E): Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Description: as for outcome 32
Time Frame: Baseline through Day 29
Population: Treatment 7-8 Amendment (C-E): No participants met the criteria (duration had to be 24 or more, and had to occur on Day 29 or before).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e))
Number analyzed (Participants) | 101 | 101
percentage of participants | 1.0 [0.0 to 2.9] | 0.0 [0.0 to 0.0]

34. Secondary Outcome: Treatment 9-11 Amendment (f), Low Risk Participants: Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Description: as for outcome 32
Time Frame: Baseline through Day 29
Population: Treatment 9-11 Amendment (f), Low Risk Participants: All participants randomly assigned and who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants)
Number analyzed (Participants) | 125 | 127 | 128
percentage of participants | 1.6 [0.0 to 3.8] | 2.4 [0.0 to 5.0] | 1.6 [0.0 to 3.7]

35. Secondary Outcome: Treatment 12 -13 Amendment (f), High Risk Participants: Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Description: as for outcome 32
Time Frame: Baseline through Day 29
Population: Treatment 12 -13 Amendment (f), High Risk Participants: All participants randomly assigned and who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants)
Number analyzed (Participants) | 100 | 50
percentage of participants | 6.0 [1.3 to 10.7] | 6.0 [0.0 to 12.6]

36. Secondary Outcome: Treatment 14 Amendment (g): Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-19 Related Emergency Room Visit, or Death From Any Cause
Description: as for outcome 32
Time Frame: Baseline through Day 29
Population: Treatment 14 Amendment (g): All participants randomly assigned and who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB(Amendment (g), High Risk,Updated CDC Criteria)
Number analyzed (Participants) | 176
percentage of participants | 2.3 [0.1 to 4.5]

37. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of Bamlanivimab
Description: PK: Mean Concentration of Bamlanivimab
Time Frame: Day 29
Population: All randomized participants who received 700 mg BAM and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter (µg/mL)
Groups:
- 700 mg BAM: Participants received 700 mg BAM administered IV.
Arm/Group | 700 mg BAM
Number analyzed (Participants) | 374
Microgram/milliliter (µg/mL) | 30.0 (36.4)

38. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of Etesevimab
Description: Pharmacokinetics (PK): Mean Concentration of Etesevimab
Time Frame: Day 29
Population: All randomized participants who received 1400 ETE and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 1400 mg ETE: Participants received 1400 mg ETE administered IV.
Arm/Group | 1400 mg ETE
Number analyzed (Participants) | 319
µg/mL | 105 (36.0)

39. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of Bebtelovimab
Description: Pharmacokinetics (PK): Mean Concentration of Bebtelovimab
Time Frame: Day 29
Population: All randomized participants who received 175 mg BEB and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 175 mg BEB: Participants received 175 mg BEB administered IV.
Arm/Group | 175 mg BEB
Number analyzed (Participants) | 520
µg/mL | 4.18 (80.4)

40. Secondary Outcome: Pharmacokinetics (PK): Mean Concentration of VIR-7831
Description: PK: Mean Concentration of VIR-7831
Time Frame: Day 29
Population: All randomized participants who received 500 mg VIR-7831 and had evaluable PK data.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 500 mg VIR-7831: Participants received 500 mg VIR-7831 administered IV.
Arm/Group | 500 mg VIR-7831
Number analyzed (Participants) | 64
µg/mL | 46.3 (47.4)

ADVERSE EVENTS:
Time Frame: Baseline Up To 169 Days
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g)), High Risk,Updated CDC Criteria): Amendment (f) High Risk Participants updated CDC criteria:
  Participants received 700 mg BAM +1400 mg ETE + 175 mg BEB administered IV.
Arm/Group | Treatment 1: Pbo | Treatment 2: 175 mg BAM +350 mg ETE | Treatment 3: 700 mg BAM +1400 mg ETE | Treatment 4: 2800 mg BAM +2800 mg ETE | Treatment 5: 700 mg BAM | Treatment 6: 350 mg BAM +700 mg ETE | Unintentional Dosing: 700 mg BAM +700 mg ETE | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g)), High Risk,Updated CDC Criteria) | 700 mg BAM 15-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) | Pooled Placebo (Addendum 4, IV) | 70 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 140 mg/Min (Addendum 4, IV) | 175 mg BEB 350 mg/Min (Addendum 4, IV) | 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) | 1750 mg BEB 350 mg/Min (Addendum 4, IV) | Pooled Placebo (Addendum 4, SC) | 280 mg BEB (Addendum 4, SC) | 560 mg BEB (Addendum 4, SC)
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/83 | 0/158 | 0/103 | 0/105 | 0/101 | 0/20 | 0/101 | 0/101 | 0/125 | 1/127 | 0/128 | 1/100 | 0/50 | 0/176 | 0/30 | 0/6 | 0/30 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/83 | 1/158 | 0/103 | 0/105 | 2/101 | 1/20 | 0/101 | 0/101 | 0/125 | 1/127 | 0/128 | 3/100 | 2/50 | 2/176 | 0/30 | 0/6 | 1/30 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 16/155 | 14/83 | 13/158 | 9/103 | 12/105 | 7/101 | 4/20 | 6/101 | 10/101 | 11/125 | 15/127 | 10/128 | 19/100 | 7/50 | 20/176 | 3/30 | 0/6 | 2/30 | 1/10 | 0/6 | 2/6 | 0/6 | 1/6 | 1/6 | 1/4 | 2/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment 1: Pbo (N=155) | Treatment 2: 175 mg BAM +350 mg ETE (N=83) | Treatment 3: 700 mg BAM +1400 mg ETE (N=158) | Treatment 4: 2800 mg BAM +2800 mg ETE (N=103) | Treatment 5: 700 mg BAM (N=105) | Treatment 6: 350 mg BAM +700 mg ETE (N=101) | Unintentional Dosing: 700 mg BAM +700 mg ETE (N=20) | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) (N=101) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) (N=101) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) (N=125) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) (N=127) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) (N=128) | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) (N=100) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) (N=50) | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g)), High Risk,Updated CDC Criteria) (N=176) | 700 mg BAM 15-min (Addendum (2)) (N=30) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) (N=6) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) (N=30) | Pooled Placebo (Addendum 4, IV) (N=10) | 70 mg BEB 140 mg/Min (Addendum 4, IV) (N=6) | 175 mg BEB 140 mg/Min (Addendum 4, IV) (N=6) | 175 mg BEB 350 mg/Min (Addendum 4, IV) (N=6) | 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) (N=6) | 1750 mg BEB 350 mg/Min (Addendum 4, IV) (N=6) | Pooled Placebo (Addendum 4, SC) (N=4) | 280 mg BEB (Addendum 4, SC) (N=6) | 560 mg BEB (Addendum 4, SC) (N=6)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 0/50 (0) | 0/48 (0) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 1/76 (1) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment 1: Pbo (N=155) | Treatment 2: 175 mg BAM +350 mg ETE (N=83) | Treatment 3: 700 mg BAM +1400 mg ETE (N=158) | Treatment 4: 2800 mg BAM +2800 mg ETE (N=103) | Treatment 5: 700 mg BAM (N=105) | Treatment 6: 350 mg BAM +700 mg ETE (N=101) | Unintentional Dosing: 700 mg BAM +700 mg ETE (N=20) | Treatment 7: 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) (N=101) | Treatment 8: Pbo For 700 mg BAM + 500 mg VIR-7831 (Amendment (C-e)) (N=101) | Treatment 9: 175 mg BEB (Amendment (f), Low Risk Participants) (N=125) | Treatment 10: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), Low Risk Participants) (N=127) | Treatment 11: Pbo For 175 mg BEB & 700 mg BAM +1400 mg ETE +175 mg BEB (Low Risk Participants) (N=128) | Treatment 12: 175 mg BEB (Amendment (f), High Risk Participants) (N=100) | Treatment 13: 700 mg BAM +1400 mg ETE +175 mg BEB (Amendment (f), High Risk Participants) (N=50) | Treatment 14: 700 mg BAM + 1400 mg ETE + 175 mg BEB (Amendment (g)), High Risk,Updated CDC Criteria) (N=176) | 700 mg BAM 15-min (Addendum (2)) (N=30) | 700 mg BAM + 1400 mg ETE 30-min (Addendum (2)) (N=6) | 700 mg BAM + 1400 mg ETE 15-min (Addendum (2)) (N=30) | Pooled Placebo (Addendum 4, IV) (N=10) | 70 mg BEB 140 mg/Min (Addendum 4, IV) (N=6) | 175 mg BEB 140 mg/Min (Addendum 4, IV) (N=6) | 175 mg BEB 350 mg/Min (Addendum 4, IV) (N=6) | 175/700/1400 mg BAM + ETE + BEB 350 mg/Min (Addendum 4, IV) (N=6) | 1750 mg BEB 350 mg/Min (Addendum 4, IV) (N=6) | Pooled Placebo (Addendum 4, SC) (N=4) | 280 mg BEB (Addendum 4, SC) (N=6) | 560 mg BEB (Addendum 4, SC) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 0/50 (0) | 0/48 (0) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 0/76 (0) | 1/72 (1) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Product administration interrupted (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood oestrogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 0/50 (0) | 1/48 (1) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 0/76 (0) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/80 (0) | 0/44 (0) | 0/72 (0) | 0/48 (0) | 0/55 (0) | 0/53 (0) | 0/12 (0) | 1/49 (1) | 0/45 (0) | 0/62 (0) | 0/51 (0) | 0/56 (0) | 0/48 (0) | 0/24 (0) | 0/78 (0) | 0/18 (0) | 0 (0) | 0/17 (0) | 0/7 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/1 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 1/50 (1) | 0/48 (0) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 0/76 (0) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 0/50 (0) | 0/48 (0) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 1/63 (1) | 0/76 (0) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 1/50 (1) | 0/48 (0) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 0/76 (0) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 0/80 (0) | 0/44 (0) | 0/72 (0) | 0/48 (0) | 0/55 (0) | 0/53 (0) | 0/12 (0) | 0/49 (0) | 0/45 (0) | 1/62 (1) | 0/51 (0) | 0/56 (0) | 0/48 (0) | 0/24 (0) | 0/78 (0) | 0/18 (0) | 0 (0) | 0/17 (0) | 0/7 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/1 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0/75 (0) | 0/39 (0) | 0/86 (0) | 0/55 (0) | 0/50 (0) | 1/48 (1) | 0/8 (0) | 0/52 (0) | 0/56 (0) | 0/63 (0) | 0/76 (0) | 0/72 (0) | 0/52 (0) | 0/26 (0) | 0/98 (0) | 0/12 (0) | 0 (0) | 0/13 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/1 (0) | 0/2 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Piloerection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: Protocol: J2X-MC-PYAH (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT04634409/Prot_000.pdf
  • Study Protocol: Protocol Addendum 2: J2X-MC-PYAH (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT04634409/Prot_001.pdf
  • Study Protocol: Protocol Addendum 4: J2X-MC-PYAH (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04634409/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04634409/SAP_003.pdf